CLINICAL TRIAL: NCT03436407
Title: Evaluation of Implementation of Pre-exposure Prophylaxis (PrEP) in Subjects at Particular Risk of Infection With Human Immunodeficiency Virus (HIV).
Brief Title: Evaluation of Implementation of Pre-exposure Prophylaxis (PrEP) in Norway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Olaug Olsen, Senior consultant/Assoc Prof, Oslo University Hospital
Other Study IDs: 2017/759
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Hiv; Sexually Transmitted Diseases; Mental Health Wellness 1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- PrEP Group: Subject offered to start PrEP treatment in routine clinical practice
- Control Group: 1. Enrolled patients will be regarded as their own control when it comes to their sexual health and quality of life reported for period prior to inclusion in the study.
  2. Subjects diagnosed with HIV within last 12 months in general clinical practice and referred to the outpatient clinic at the Dept. of Infectious Diseases, OUS. (details in protocol 3.3.2)
  3. Frequency of STI reported to the National Institute of Public Health (MSIS) will be compared with the frequency of STIs in the study cohort.

SUMMARY:
Despite the significant preventive efforts to reduce HIV infections in the past decades, the incidence in MSM has plateaued at a higher level after the turn of the millennium. In 2015 a reduction in newly diagnosed HIV cases was reported for the first time. Early detection of HIV and treatment as prevention may have played a positive role in reducing HIV transmission, however, numbers increased again in 2016. Over 90% of HIV positive MSM in Norway are treated and virologically suppressed and thereby considered not infectious.

Since the early days of the HIV epidemic, changes in sexual behaviour and increased use of condoms have been advocated and the only tools available to prevent HIV transmission. Later, frequent testing and treatment of STIs (including HIV) have been added to the preventive measures available. Still, this does not seem to be sufficient for all MSM. The use of PrEP is therefore likely an important supplement to prevent HIV infections in MSM at high risk for HIV acquisition.

The main objective of this study is to monitor the impact of PrEP on the subject's psychological and sexual health. It is also important to monitor the adherence to PrEP, development of drug resistance (in the case of undetected HIV infection at initiation of PrEP), frequency of other STIs, changes in sexual behaviour, recreational drug use and quality of life. PrEP has proven to be effective in reducing the sexual acquisition of HIV, however this requires that the medication is taken as prescribed, whilst the subject is exposed to high risk of infection.

DETAILED DESCRIPTION:
This study is designed to evaluated implementation of PrEP treatment as a part of the general HIV preventive program in Norway. The target groups are mainly MSM and transgender persons at high risk of HIV infection, as well as other subjects at risk of HIV infection due to their sexual practices.

Objectives include assessment of the following:

1. Assess the impact of PrEP on the sexual and psychological health of PrEP users Incidence of sexually transmitted infections (STIs) in PrEP users compared to those not taking PrEP
2. Assessment of drug compliance
3. Incidence of HIV seroconversion despite PrEP
4. Frequency and development of drug resistance in subjects who HIV-seroconvert (if any)

ELIGIBILITY:
Inclusion Criteria:

1. Male, female or transgender persons aged ≥ 18 years who are offered or have started PrEP in routine clinical practice, and 2, 3, 4, 5, 6 or 7 (below).
2. Men who have sex with men (MSM) and transgender persons;

   1. who have had unprotected anal sex with two or more partners during the last six months and/or
   2. who have had bacterial sexually transmittable infection(s) during the last twelve months and/or
   3. who have used post-exposure prophylaxis(PEP) during the last twelve months and/or
   4. who use recreational drugs when having sex
3. Indication for PrEP is present according to the assessment of the health care provider
4. Men and women who are at high risk of HIV according to their sexual practices
5. HIV-negative partner of a HIV-positive person not yet virologically suppressed by antiretroviral therapy (ART)
6. Sex workers with inconsistent condom use
7. Persons with inconsistent condom use with sexual partners in / from countries with a high prevalence of HIV (COHP)

Exclusion Criteria:

1. HIV positive subjects
2. Subjects who cannot take Emtricitabine/tenofovir disoproxil combination tablet (FTC/TDF) due to contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender
Study Population: Individuals attending the clinic for PrEP assessment are either referred from other health care providers or referred by themselves (self-referral).
  Those who have commenced PrEP elsewhere (abroad, purchased themselves, another provider) and attend for "PrEP follow-up" either at Olafiaklinikken or a corresponding venerological clinic/study site in Norway, may also be included in the study.
  Newly diagnosed HIV positive individuals referred to the out-patient clinic of the Dept. of Infectious Diseases, OUS, will be invited to participate as controls. They will be presented with the same consent form and questionnaire on sexual and psychological health prior to the HIV diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of PrEP | 24 months
  Assess the impact of PrEP on the sexual and psychological health of PrEP users

SECONDARY OUTCOMES:
Incidence of STIs | 24 months
  Incidence of sexually transmitted infections (STIs) in PrEP users compared to those not taking PrEP
Drug compliance | 24 months
  Assessment of drug compliance
HIV seroconversion | 24 months
  Incidence of HIV seroconversion despite PrEP
Drug resistance | 24 months
  Frequency and development of drug resistance in subjects who HIV-seroconvert

CONTACTS AND LOCATIONS:
Overall Officials: Anne Olaug Olsen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (9):
- Norway (9):
  - Helse Bergen HF - Haukeland universitetssykehus, Bergen
  - Sørlandet sykehus HF, Kristiansand
  - Olafia Clinic,Oslo University Hosptial, Oslo
  - Akershus universitetssykehus HF, Oslo
  - Brynsenglegene, Oslo
  - Dept. Inf. Diseases, Oslo University Hospital, Oslo
  - Helse Stavanger HF - Stavanger universitetssjukehus, Stavanger
  - Universitetssykehuset Nord-Norge HF, Tromsø
  - Helse Midt-Norge St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03436407/SAP_000.pdf
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT03436407/Prot_001.pdf
  • Informed Consent Form (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT03436407/ICF_002.pdf